CLINICAL TRIAL: NCT04664959
Title: A Phase III, Randomised, Double-blind, Multicentre Clinical Study to Compare the Efficacy, Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity Between SB16 (Proposed Denosumab Biosimilar) and Prolia® in Postmenopausal Women With Osteoporosis
Brief Title: A Study to Compare SB16 (Proposed Denosumab Biosimilar) to Prolia® in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB16-3001
Record Dates: First submitted 2020-12-10; First posted 2020-12-11 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SB16 (Proposed Denosumab Biosimilar) (Experimental): Subjects randomised into SB16 group will receive SB16 (60 mg in 1 mL) subcutaneously every 6 months.
  Interventions: Drug: SB16 (Proposed Denosumab Biosimilar)
- Prolia® (Denosumab) (Active Comparator): Subjects randomised into Prolia® group will receive Prolia® (60 mg in 1 mL) subcutaneously every 6 months.
  At Month 12, subjects in Prolia® treatment group will be re-randomised in a 1:1 ratio to either continue on Prolia® treatment or be transitioned to SB16 treatment. After re-randomisation, subjects transited to SB16 group will receive SB16, and subjects remaining in Prolia® group will continue to receive Prolia® at Month 12.
  Interventions: Drug: SB16 (Proposed Denosumab Biosimilar); Drug: Prolia® (Denosumab)

INTERVENTIONS:
Drug: SB16 (Proposed Denosumab Biosimilar) — Subjects randomised into SB16 group will receive SB16 (60 mg in 1 mL) subcutaneously every 6 months.
  At Month 12, subjects transited from Prolia® group to SB16 group will receive SB16 (60 mg in 1 mL) subcutaneously.
Drug: Prolia® (Denosumab) — Subjects randomised into Prolia® group will receive Prolia® (60 mg in 1 mL) subcutaneously every 6 months.
  Arms: Prolia® (Denosumab)

SUMMARY:
This is a randomised, double-blind, multicentre study to evaluate the efficacy, safety, PK, PD, and immunogenicity of SB16 compared to Prolia® in postmenopausal women with osteoporosis.

DETAILED DESCRIPTION:
Subjects will be randomised in a 1:1 ratio to receive either SB16 or Prolia®. At Month 12, subjects in Prolia® treatment group will be randomised again in a 1:1 ratio to either continue on Prolia® treatment or be transitioned to SB16 treatment. Investigational product (60 mg in 1 mL of SB16 or Prolia®) will be given subcutaneously every 6 months up to Month 12, and the last assessment will be done at Month 18.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women who are 55 to 80 years of age at Screening
* Ambulatory and visually unimpaired to participate in the study at Screening, in the opinion of the Investigator
* Absolute BMD consistent with T-score at the total hip or lumbar spine of -4 and -2.5 at Screening
* At least three evaluable vertebrae within L1 to L4, one evaluable femoral neck, and one evaluable hip joint for BMD measurement at Screening
* Biologic naïve at Screening
* Body weight of 50 kg and 90 kg at Screening

Exclusion Criteria:

* One severe or more than two moderate vertebral fractures on spinal X-ray according to Genant classification at Screening
* History of hip fracture or bilateral hip replacement at Screening
* Uncorrected vitamin D deficiency at Screening
* Hypercalcemia or hypocalcaemia at Screening
* Inadequate haematological function at Screening
* Inadequate renal or hepatic function at Screening
* Known allergic reactions, hypersensitivity, or intolerance to denosumab or to any ingredients of the IP, including latex allergy or hereditary problems of fructose intolerance at Screening
* May not tolerate long-term calcium or vitamin D supplementation or subject with malabsorption of calcium or vitamin D supplements, in the opinion of the Investigator, at Screening
* Use of any of the medications that can affect BMD
* Use of any non-biologic IP that is not indicated for osteoporosis from another study or use of an investigational device at Screening
* Non-osteoporosis medical conditions that can affect BMD at Screening
* Any clinically significant disease or disorder or laboratory abnormality which, in the opinion of the Investigator, would prevent the subject from completing the study or the interpretation of the study results at Screening and Randomisation

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2023-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Poland (5):
  - SB Investigative Site, Krakow
  - SB Investigative Site, Lodz
  - SB Investigative Site, Siedlce
  - SB Investigative Site, Warsaw
  - SB Investigative Site, Zamość

REFERENCES:
- [Derived] Langdahl B, Chung YS, Plebanski R, Czerwinski E, Dokoupilova E, Supronik J, Rosa J, Mydlak A, Rowinska-Osuch A, Baek KH, Urboniene A, Mordaka R, Ahn S, Rho YH, Ban J, Eastell R. Proposed Denosumab Biosimilar SB16 vs Reference Denosumab in Postmenopausal Osteoporosis: Phase 3 Results Up to Month 12. J Clin Endocrinol Metab. 2025 May 19;110(6):e1951-e1958. doi: 10.1210/clinem/dgae611. PMID 39243386

RESULTS

PARTICIPANT FLOW:
Groups:
- SB16: Subjects were randomly assigned to receive SB16 subcutaneously 60 mg at Months 0 and 6.
- Prolia: Subjects were randomly assigned to receive Prolia subcutaneously 60 mg at Months 0 and 6.
- SB16+SB16: Subjects were randomly assigned to receive SB16 subcutaneously 60 mg at Months 0 and 6. At Month 12, subjects who received SB16 in the Main period continued to receive SB16, but they also followed the randomisation procedure to maintain blinding.
- Prolia+SB16; Prolia+Prolia: Subjects were randomly assigned to receive Prolia subcutaneously 60 mg at Months 0 and 6. At Month 12, subjects who received Prolia in the Main period of the SB16-3001 study were randomised again in a 1:1 ratio to either continue on Prolia (Prolia+Prolia) or were transitioned to SB16 (Prolia+SB16).
Period: Main Period
Arm/Group | SB16 | Prolia | SB16+SB16 | Prolia+SB16 | Prolia+Prolia
Started | 225 | 232 | 0 | 0 | 0
Completed | 206 | 201 | 0 | 0 | 0
Not Completed | 19 | 31 | 0 | 0 | 0
Period: Transition Period
Arm/Group | SB16 | Prolia | SB16+SB16 | Prolia+SB16 | Prolia+Prolia
Started | 0 | 0 | 206 | 100 | 101
Completed | 0 | 0 | 206 | 99 | 99
Not Completed | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB16 | Prolia | Total
Number analyzed (Participants) | 225 | 232 | 457
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 95 | 184
  >=65 years | 136 | 137 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (5.87) | 66.3 (6.03) | 66.4 (5.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 225 | 232 | 457
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 18 | 23 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 207 | 208 | 415
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 12
Time Frame: Baseline and Month 12
Measure: Least Squares Mean (Standard Error); unit: %Change of BMD
Arm/Group | SB16 | Prolia
Number analyzed (Participants) | 225 | 231
%Change of BMD | 5.63 (0.250) | 5.30 (0.254)

ADVERSE EVENTS:
Time Frame: Overall Period (18 months)
Groups:
- SB16: Subjects were randomly assigned to receive SB16 subcutaneously 60 mg at Months 0 and 6. At Month 12, subjects who received SB16 in the Main period continued to receive SB16, but they also followed the randomisation procedure to maintain blinding.
- Prolia Overall: Prolia Overall include subjects who had randomised to Prolia at Month 0 and had re-randomisation (Prolia+SB16 or Prolia+Prolia) at Month 12. Prolia+SB16 and Prolia+Prolia may not add up to Prolia Overall.
Arm/Group | SB16 | Prolia Overall | Prolia+SB16 | Prolia+Prolia
All-Cause Mortality (participants affected / at risk) | 0/225 | 0/231 | 0/100 | 0/101
Serious Adverse Events (participants affected / at risk) | 12/225 | 11/231 | 5/100 | 3/101
Other Adverse Events (participants affected / at risk) | 116/225 | 107/231 | 46/100 | 49/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SB16 (N=225) | Prolia Overall (N=231) | Prolia+SB16 (N=100) | Prolia+Prolia (N=101)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 0
Urethral caruncle (Renal and urinary disorders) | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SB16 (N=225) | Prolia Overall (N=231) | Prolia+SB16 (N=100) | Prolia+Prolia (N=101)
Headache (Nervous system disorders) | 17 | 13 | 8 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 12 | 7 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 | 11 | 5 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 6 | 0
COVID-19 (Infections and infestations) | 20 | 18 | 5 | 11
Upper respiratory tract infection (Infections and infestations) | 13 | 12 | 3 | 5
Urinary tract infection (Infections and infestations) | 13 | 7 | 1 | 5
Nasopharyngitis (Infections and infestations) | 10 | 18 | 7 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 23 | 27 | 11 | 13
Hypercholesterolaemia (Metabolism and nutrition disorders) | 16 | 7 | 2 | 5
Vitamin D deficiency (Metabolism and nutrition disorders) | 11 | 9 | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT04664959/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT04664959/SAP_001.pdf